CLINICAL TRIAL: NCT03603600
Title: A Prospective, Multicenter, Randomized, Active-Controlled Clinical Study to Evaluate the Safety and Effectiveness of the enVista® One-Piece Hydrophobic Acrylic Trifocal Intraocular Lens in Subjects Undergoing Cataract Extraction
Brief Title: Evaluate the Safety and Effectiveness of the enVista® One-Piece Hydrophobic Acrylic Trifocal Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 945
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Approximately 334 subjects will be implanted bilaterally with the enVista MX60EF trifocal MIOL, and approximately 167 control subjects will be implanted bilaterally with the enVista MX60E monofocal IOL
Who Masked: Participant, Outcomes Assessor
Masking Description: The Investigator implanting the IOL and designated site personnel will be unmasked to the assignment of IOLs. Subjects and designated postoperative evaluator(s) will be masked to the IOLs assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- enVista MX60EF (Experimental): enVista MX60EF (trifocal) multifocal IOL (MIOL)
  Interventions: Device: enVista MX60EF
- enVista MX60E (Active Comparator): enVista MX60E monofocal IOL
  Interventions: Device: enVista MX60E

INTERVENTIONS:
Device: enVista MX60E — enVista MX60E monofocal IOL
  Arms: enVista MX60E
Device: enVista MX60EF — enVista MX60EF (trifocal) multifocal IOL (MIOL)
  Arms: enVista MX60EF

SUMMARY:
The objective of the study is to evaluate the safety and effectiveness of the enVista trifocal intraocular lens when implanted in the capsular bag.

DETAILED DESCRIPTION:
Cataracts are a common condition in adults over 40 years of age, and surgical replacement of the cataractous lens with an intraocular lens (IOL) remains an effective way to restore vision to cataract patients.The objective of the study is to evaluate the safety and effectiveness of the enVista trifocal intraocular lens when implanted in the capsular bag.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 22 years of age or older on the date the Informed Consent Form (ICF) is signed.
2. Subjects must have the capability to understand and provide written informed consent on the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved Informed Consent Form (ICF) and authorization as appropriate for local privacy regulations.
3. Subjects must have a BCDVA equal to or worse than 20/40 in each eye, with or without a glare source, due to a clinically significant cataract (cortical, nuclear, subcapsular, or combination) that is considered amenable to treatment with standard phacoemulsification cataract extraction and capsular IOL implantation.
4. Subjects must have a BCDVA projected to be better than 20/32 after IOL implantation in each eye, as determined by the medical judgment of the Investigator or measured by potential acuity meter (PAM) testing, if necessary.
5. Subjects must have clear intraocular media other than the cataract in both eyes.
6. Contact lens wearers must demonstrate a stable refraction (within ±0.50 D for both sphere and cylinder) in both eyes, as determined by distance manifest refraction on two consecutive examination dates after discontinuation of contact lens wear.
7. Subjects must require an IOL power from +16.0 diopter (D) to +24.0 D in both eyes.
8. Subjects must be willing and able to comply with all treatment and follow-up study visits and procedures, and to undergo second eye surgery within 7-30 days of the first eye surgery.

Exclusion Criteria:

1. Subjects who have used an investigational drug or device within 30 days prior to entry into this study and/or will participate in another investigation during the period of study participation.
2. Subjects who have any corneal pathology (e.g., significant scarring, guttata, inflammation, edema, dystrophy, etc.) in either eye.
3. Subjects who have significant anterior segment pathology that might increase intraoperative risk or compromise IOL stability (e.g., pseudoexfoliation syndrome, synechiae, iris atrophy, traumatic cataract, lens subluxation, traumatic zonulolysis, zonular dialysis, evident zonular weakness or dehiscence, hypermature or brunescent cataract, etc.) in either eye.
4. Subjects who have uncontrolled glaucoma in either eye.
5. Subjects who have previous retinal detachment or clinically significant retinal pathology involving the macula in either eye.
6. Subjects who have proliferative or non-proliferative diabetic retinopathy in either eye.
7. Subjects who have a congenital ocular anomaly (e.g., aniridia, congenital cataract) in either eye.
8. Subjects using any systemic or topical drug known to interfere with visual performance, pupil dilation, or iris structure within 30 days of enrollment or during the study (refer to the relevant attachment of the Study Reference Manual).
9. Subjects who have a history of chronic or recurrent inflammatory eye disease (e.g., iritis, scleritis, iridocyclitis, or rubeosis iridis) in either eye.
10. Subjects who have a visual disorder, other than cataracts, that could potentially cause future acuity losses to a level of 20/100 or worse in either eye.
11. Subjects who have had previous intraocular or corneal surgery in either eye, with the exception of laser trabeculoplasty.
12. Subjects with any preoperative infectious conjunctivitis, keratitis, or uveitis in either eye.
13. Subjects who have a preoperative corneal astigmatism > 1.0 D in either eye, irregular astigmatism, or skewed radial axis (note: corneal incisions intended specifically to reduce astigmatism are not allowed during the study).
14. Subjects who cannot achieve a minimum pharmacologic pupil dilation of 5.0 mm in both eyes.
15. Subjects who may be expected to require a combined or other secondary surgical procedure in either eye.
16. Subjects who during the first cataract extraction experience an anterior or posterior capsule tear or rupture, zonular dialysis, significant iris trauma, or other complication that may cause untoward effects in the judgment of the Investigator.
17. Females of childbearing potential (those who are not surgically sterilized or at least 12 months postmenopausal) are excluded from enrollment in the study if they are currently pregnant or plan to become pregnant during the study. Females of childbearing potential must be willing to practice effective contraception for the duration of the study.
18. Subjects with any other serious ocular pathology or underlying systemic medical condition (e.g., uncontrolled diabetes) or circumstance that, based on the Investigator's judgment, poses a concern for the subjects' safety or could confound the results of the study.
19. Subjects who have current or previous usage of an alpha-1-selective adrenoceptor blocking agent or an antagonist of alpha 1A adrenoceptor (e.g., Flomax® (tamsulosin HCl), Terazosin, or Cardura).

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosangela Nolasco, Study Director — Bausch & Lomb Incorporated
Locations (23):
- United States (23):
  - Bausch Site 108, Fayetteville, Arkansas
  - Bausch Site 113, Garden Grove, California
  - Bausch Site 120, Northridge, California
  - Bausch Site 115, Redding, California
  - Bausch Site 103, Torrance, California
  - Bausch Site 107, Mt. Dora, Florida
  - Bausch Site 117, Lake Villa, Illinois
  - Bausch Site 101, Bloomington, Minnesota
  - Bausch Site 119, Birmingham, Mississippi
  - Bausch Site 102, St Louis, Missouri
  - Bausch Site 124, Omaha, Nebraska
  - Bausch Site 118, Las Vegas, Nevada
  - Bausch Site 106, Brecksville, Ohio
  - Bausch Site 109, Columbus, Ohio
  - Bausch Site 116, Pittsburgh, Pennsylvania
  - Bausch Site 121, Sioux Falls, South Dakota
  - Bausch Site 112, Memphis, Tennessee
  - Bausch Site 110, Nashville, Tennessee
  - Bausch Site 104, Cedar Park, Texas
  - Bausch Site 105, Dallas, Texas
  - Bausch Site 111, Houston, Texas
  - Bausch Site 122, San Antonio, Texas
  - Bausch Site 123, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | enVista MX60EF | enVista MX60E
Started | 332 | 169
Completed | 319 | 157
Not Completed | 13 | 12
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Lost to Follow-up | 2 | 3
Not completed — Death | 3 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Other reason | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | enVista MX60EF | enVista MX60E | Total
Number analyzed (Participants) | 332 | 169 | 501
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (7.89) | 68.8 (7.46) | 68.0 (7.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 108 | 320
  Male | 120 | 61 | 181
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 20 | 60
  Not Hispanic or Latino | 292 | 149 | 441
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 4 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 14 | 9 | 23
  White | 305 | 156 | 461
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 322 | 169 | 501

OUTCOME MEASURES:

1. Primary Outcome: Photopic Monocular Best-corrected Distance Visual Acuity (BCDVA)
Description: Photopic monocular best-corrected distance visual acuity (BCDVA) in first eyes at Post-Operative Visit 4 (Day 120 to 180 after second eye implantation eyes at Post-Operative Visit 4 (Day 120 to 180 after second eye implantation)
Time Frame: Day 120 to Day 180 after second eye implantation, up to 210 days from first eye implantation at Baseline.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | enVista MX60EF | enVista MX60E
Number analyzed (Participants) | 312 | 156
logMAR | 0.022 (0.0950) | -0.017 (0.0897)

2. Primary Outcome: Photopic Monocular Distance-corrected Near Visual Acuity (DCNVA)
Description: Photopic monocular distance-corrected near visual acuity (DCNVA) in first eyes at 40 cm at Post-Operative Visit 4 (Day 120 to 180 after second eye IOL implantation)
Time Frame: Day 120 to Day 180 after second eye implantation, up to 210 days from first eye implantation at Baseline.
Population: Modified Intent to Treat Set Excluding Phase I Subjects
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | enVista MX60EF | enVista MX60E
Number analyzed (Participants) | 297 | 152
logMAR | 0.152 (0.1342) | 0.545 (0.1703)

3. Primary Outcome: Photopic Monocular Distance-corrected Intermediate Visual Acuity (DCIVA)
Description: Photopic monocular distance-corrected intermediate visual acuity (DCIVA) in first eyes at 66 cm at Post-Operative Visit 4 (Day 120 to 180 after second eye IOL implantation
Time Frame: Day 120 to Day 180 after second eye implantation, up to 210 days from first eye implantation at Baseline.
Population: Modified Intent to Treat Set Excluding Phase I Subjects
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | enVista MX60EF | enVista MX60E
Number analyzed (Participants) | 297 | 152
logMAR | 0.122 (0.1199) | 0.349 (0.1592)

4. Primary Outcome: Serious Adverse Events
Description: All ocular SAEs, including secondary surgical interventions (SSIs) related to the optical properties of the IOL, in first eyes through study exit
Time Frame: Assessed through study exit, 330 - 450 days after second eye implantation, up to 480 days from first eye implantation at baseline
Population: Modified Safety Set: The Modified Safety Set included all subjects with at least 1 eye in which the IOL touched the eye with a study lens.
Measure: Count of Participants; unit: Participants
Arm/Group | enVista MX60EF | enVista MX60E
Number analyzed (Participants) | 332 | 169
Participants
  Macular hole | 1 | 0
  Retinal tear | 1 | 0
  Retinal vein occlusion | 1 | 0
  Ophthalmic herpes zoster | 0 | 1
  Seidel test positive | 1 | 0

5. Primary Outcome: The Rate of SSIs Due to the Optical Properties of the Lens for First Eyes Through Study Exit
Description: The cumulative rate of secondary surgical interventions (SSI) due to the optical properties of the lens for first eyes through study exit. The rate was determined as the number of first eyes with an SSI related to the optical properties of the IOL divided by the total number of first eyes.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: first eyes
Arm/Group | enVista MX60EF | enVista MX60E
Number analyzed (Participants) | 332 | 169
first eyes | 0 | 0

6. Primary Outcome: The Incidence of AEs in First Eyes Compared to ISO Safety and Performance Endpoint
Description: as for outcome 5
Time Frame: as for outcome 4
Population: The measure was not assessed for the control arm.
Measure: Number; unit: first eyes
Arm/Group | enVista MX60EF
Number analyzed (Participants) | 332
first eyes
  Cystoid macular oedema | 0
  Hypopyon | 0
  Endophthalmitis | 0
  Lens dislocated from posterior chamber | 0
  Pupillary block | 0
  Retinal detachment | 0
  SSI | 0

7. Secondary Outcome: Photopic Binocular DCNVA at 40 cm at Postoperative Visit 4
Description: Photopic binocular distance-corrected near visual acuity (DCNVA) at 40 cm at Post-Operative Visit 4 (Day 120 to 180 after second eye IOL implantation)
Time Frame: Day 120 to Day 180 after second eye implantation, up to 210 days from first eye implantation at Baseline.
Population: Modified Intent to Treat Set Excluding Phase I Subjects
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | enVista MX60EF | enVista MX60E
Number analyzed (Participants) | 284 | 142
logMAR | 0.080 (0.0977) | 0.453 (0.1526)

8. Secondary Outcome: Photopic Binocular UNVA at 40 cm at Postoperative Visit 4
Description: Photopic binocular uncorrected near visual acuity (UNVA) at 40 cm at Post-Operative Visit 4 (Day 120 to 180 after second eye IOL implantation)
Time Frame: Day 120 to Day 180 after second eye implantation, up to 210 days from first eye implantation at Baseline.
Population: Modified Intent to Treat Set Excluding Phase I Subjects
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | enVista MX60EF | enVista MX60E
Number analyzed (Participants) | 297 | 153
logMAR | 0.096 (0.1056) | 0.418 (0.1454)

9. Secondary Outcome: Photopic Binocular DCIVA at 66 cm at Postoperative Visit 4
Description: Photopic binocular distance-corrected intermediate visual acuity (DCIVA) at 66 cm at Post-Operative Visit 4 (Day 120 to 180 after second eye IOL implantation)
Time Frame: Day 120 to Day 180 after second eye implantation, up to 210 days from first eye implantation at Baseline.
Population: Modified Intent to Treat Set Excluding Phase I Subjects
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | enVista MX60EF | enVista MX60E
Number analyzed (Participants) | 283 | 142
logMAR | 0.041 (0.0976) | 0.268 (0.1485)

10. Secondary Outcome: Photopic Binocular UIVA at 66 cm at Postoperative Visit 4
Description: Photopic binocular uncorrected intermediate visual acuity (UIVA) at 66 cm at Postoperative Visit 4 (Day 120 to Day 180 after second eye implantation)
Time Frame: Day 120 to Day 180 after second eye implantation, up to 210 days from first eye implantation at Baseline.
Population: Modified Intent to Treat Set Excluding Phase I Subjects
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | enVista MX60EF | enVista MX60E
Number analyzed (Participants) | 297 | 153
logMAR | 0.064 (0.0988) | 0.217 (0.1442)

11. Secondary Outcome: First-eye BCDVA Evaluated at Postoperative Visit 5
Description: First-eye BCDVA evaluated at Postoperative Visit 5 (Day 330 to Day 420 after second eye implantation)
Time Frame: Day 330 to Day 420 after second eye implantation, up to 450 days from first eye implantation at baseline
Population: Modified Intent to Treat Set
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | enVista MX60EF | enVista MX60E
Number analyzed (Participants) | 308 | 152
logMAR | 0.027 (0.0920) | -0.020 (0.0826)

12. Secondary Outcome: First-eye DCNVA Evaluated at Postoperative Visit 5
Description: First-eye DCNVA evaluated at Postoperative Visit 5 (Day 330 to Day 420 after second eye implantation)
Time Frame: Day 330 to Day 420 after second eye implantation, up to 450 days from first eye implantation at baseline
Population: Modified Intent to Treat Set Excluding Phase I Subjects
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | enVista MX60EF | enVista MX60E
Number analyzed (Participants) | 280 | 139
logMAR | 0.143 (0.1284) | 0.533 (0.1843)

13. Secondary Outcome: First-eye DCIVA Evaluated at Postoperative Visit 5
Description: First-eye DCIVA evaluated at Postoperative Visit 5 (Day 330 to Day 420 after second eye implantation)
Time Frame: Day 330 to Day 420 after second eye implantation, up to 450 days from first eye implantation at baseline
Population: Modified Intent to Treat Set Excluding Phase I Subjects
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | enVista MX60EF | enVista MX60E
Number analyzed (Participants) | 280 | 139
logMAR | 0.120 (0.1147) | 0.343 (0.1594)

ADVERSE EVENTS:
Time Frame: Through study completion, 330 - 450 days after second eye implantation, up to 480 days from first eye implantation at baseline
Description: Ocular Adverse Events
Groups:
- enVista MX60EF: enVista MX60EF (trifocal) multifocal IOL (MIOL) Subjects implanted with enVista MX60EF trifocal intraocular lenses (IOLs). For ocular AEs, the number of eyes at risk were 661 for the enVista MX60EF trifocal intraocular lens (IOL) group
- enVista MX60E: enVista MX60E monofocal IOL Subjects implanted with enVista MX60E monofocal intraocular lenses (IOLs). For ocular AEs, the number of eyes at risk were 337 for the enVista MX60E monofocal intraocular lens (IOL) group.
Arm/Group | enVista MX60EF | enVista MX60E
All-Cause Mortality (participants affected / at risk) | 3/332 | 1/169
Serious Adverse Events (participants affected / at risk) | 17/332 | 15/169
Other Adverse Events (participants affected / at risk) | 120/332 | 47/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | enVista MX60EF (N=332) | enVista MX60E (N=169)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seidel test positive (Investigations) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 2 (2)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2)
Multiple organ dysfunction syndrome (Eye disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | enVista MX60EF (N=332) | enVista MX60E (N=169)
Punctate keratitis (Eye disorders) | 57 (57) | 16 (16)
Intraocular pressure increased (Investigations) | 43 (43) | 21 (21)
Vitreous detachment (Eye disorders) | 32 (32) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact Sponsor directly for details

DOCUMENTS (2):
  • Study Protocol (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT03603600/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT03603600/SAP_001.pdf